CLINICAL TRIAL: NCT03766854
Title: A Multiple-dose Trial Investigating the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of NNC0148-0287 C (Insulin 287) for Subcutaneous Administration in Japanese Subjects With Type 1 Diabetes
Brief Title: A Research Study of How Different Amounts of a New Medicine NNC0148-0287 C (Insulin 287) Works on the Blood Sugar of People Who Are Japanese With Type 1 Diabetes When Given Once a Week
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NN1436-4422; U1111-1211-7635 (Other: World Health Organization (WHO))
Record Dates: First submitted 2018-12-04; First posted 2018-12-06 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — insulin icodec

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Insulin 287 followed by insulin glargine U100 (Experimental): Run-in period (2 days to 7 weeks): The basal insulin glargine dose for each subject will be established and optimised.
  After run-in, participants will receive insulin 287 once a week (OW) for 8 weeks and subsequent 4 weeks of terminal pharmacokinetic (PK) sampling where subjects are treated with once daily (OD) insulin glargine.
  After insulin 287 treatment, participants will receive insulin glargine U100 OD for 2 weeks.
  Interventions: Drug: insulin icodec; Drug: Insulin glargine U100
- Insulin glargine U100 followed by insulin 287 (Experimental): Run-in period (2 days to 7 weeks): The basal insulin glargine dose for each subject will be established and optimised.
  After run-in, participants will receive insulin glargine U100 OD for 2 weeks followed by 1-14 days (at least 1 day is mandatory) of continued insulin glargine treatment.
  After insulin glargine treatment, participants will receive insulin 287 OW for 8 weeks and subsequent 4 weeks of terminal PK sampling.
  Interventions: Drug: insulin icodec; Drug: Insulin glargine U100

INTERVENTIONS:
Drug: insulin icodec — Participants will receive subcutaneous (s.c.) injections of insulin 287 once weekly for 8 weeks
  Other Names: Insulin 287
Drug: Insulin glargine U100 — Participants will receive s.c. injections of insulin glargine once weekly for 2 weeks

SUMMARY:
This study will look at how insulin 287 works, if it is safe and the side effects in people who are Japanese with type 1 diabetes. The study will test how insulin goes through your blood, how long it stays there and how the blood sugar is lowered. Insulin 287 is a new medicine. Insulin glargine is already approved to treat diabetes. The study doctors can prescribe insulin glargine. The participants will get both of the insulins in a random order. The participants will get 8 weekly doses of insulin 287 and 14 daily doses of insulin glargine. There will also be a run-in period of 2 days to 7 weeks when the participants inject insulin glargine every day before they start insulin 287 period or insulin glargine period. All doses will be injected under the skin. During the run-in period, the participants adjust the insulin glargine dose and make their blood sugar levels stable. From the run-in period, the participants will take insulin aspart as bolus insulin. The study will last for about 16 - 28 weeks. The participants will have 24 visits with the study doctor. There will be 3 glucose clamps where the participants' blood sugar is tested over time. The participants cannot be in the study if the study doctor thinks that there are risks for their health.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, Japanese subjects, aged 20 - 64 years (both inclusive) at the time of signing informed consent.
* Diagnosed with type 1 diabetes mellitus greater than or equal to 1 year prior to the day of screening.
* Current daily basal insulin treatment greater than or equal to 0.2 U/kg/day.
* Body mass index between 18.5 and 28.0 kg/m^2 (both inclusive).
* HbA1c less than or equal to 9.0%.

Exclusion Criteria:

* History or presence of any clinically relevant respiratory, metabolic, renal, hepatic, gastrointestinal or endocrinological conditions (except conditions associated with diabetes mellitus).
* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using adequate contraceptive methods.
* Known or suspected hypersensitivity to trial products or related products

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-12-07 (Actual); Primary Completion 2019-12-09 (Actual); Study Completion 2019-12-09 (Actual)

PRIMARY OUTCOMES:
AUCI287τ,SS - Area under the serum insulin 287 concentration-time curve during one dosing interval at steady state | From 0 to 168 hours after trial product administration (day 50)
  Measured in pmol*h/L

SECONDARY OUTCOMES:
Number of adverse events (AEs) | From first trial product administration (day 1) to end of last dosing interval (day 57 for insulin 287, day 15 for IGlar)
  Number of events
Number of hypoglycaemic episodes | From first trial product administration (day 1) to end of last dosing interval (day 57 for insulin 287, day 15 for IGlar) excluding clamp days
  Number of episodes
Change in antiinsulin 287 antibody level | From first insulin 287 administration (day 1) to follow-up visit (day 106)
  Measured in % B/T (percentage of bound tracer measured after precipitation to total tracer)
Change in antiinsulin 287 antibody titres | From first insulin 287 administration (day 1) to follow-up visit (day 106)
  Number of dilutions.
  The antibody titer is calculated by diluting the blood serum sample containing antibody in serial ratios (1:2, 1:4, 1:8, 1:16... and so on). Using an appropriate detection method (e.g., colorimetric, chromatographic, etc.), each dilution is tested for the presence of detectable levels of antibody. The assigned titer value is indicative of the last dilution in which the antibody was detected.
Positive cross-reactive anti-human insulin antibodies | At follow-up visit (day 106)
  Yes/no. Number of participants who developed/not developed positive cross-reactive anti-human insulin antibodies.
AUCI287,0-168,FD - Area under the serum insulin 287 concentration-time curve after the first dose | From 0 to 168 hours after trial product administration (day 1)
  Measured in pmol*h/L
tmax,I287,FD - Time to maximum observed serum insulin 287 concentration after the first dose | From 0 to 168 hours after trial product administration (day 1)
  Measured in hours
Cmax,I287,FD - Maximum observed serum insulin 287 concentration after the first dose | From 0 to 168 hours after trial product administration (day 1)
  Measured in pmol/L
tmax,I287,SS - Time to maximum observed serum insulin 287 concentration after the last dose | From 0 to 168 hours after trial product administration (day 50)
  Measured in hours
Cmax,I287,SS - Maximum observed serum insulin 287 concentration after the last dose | From 0 to 168 hours after trial product administration (day 50)
  Measured in pmol/L
t1/2,I287,SS - Terminal half-life for insulin 287 at steady state | Terminal part of the serum insulin 287 concentration-time curve where the curve is well approximated by a straight line on logarithmic scale after last trial product administration (day 50)
  Measured in hours
CI287,trough - Serum insulin 287 trough concentration | Measured at the end of each dosing interval 168 hours after dosing (day 8, 15, 22, 29, 36, 43, 50 and 57)
  Measured in pmol/L
AUCIGlar,τ,SS - Area under the serum IGlar concentration-time curve during one dosing interval at steady state | From 0 to 24 hours after trial product administration (day 14)
  Measured in pmol*h/L
Cmax,IGlar,SS - Maximum observed serum IGlar concentration at steady state | From 0 to 24 hours after trial product administration (day 14)
  Measured in pmol/L
tmax,IGlar,SS - Time to maximum observed serum IGlar concentration at steady state | From 0 to 24 hours from trial product administration (day 14)
  Measured in hours
CIGlar,trough - Serum IGlar trough concentration | Measured at the end of each dosing interval 24 hours after trial product administration (day 7, 14 and 15)
  Measured in pmol/L
AUCGIR,24-48h,SS - Area under the glucose infusion rate-time curve at steady state | From 24 to 48 hours after trial product administration (day 51)
  Measured in mg/kg
GIRmax,24-48h, SS - Maximum observed glucose infusion rate at steady state | From 24 to 48 hours after trial product administration (day 51)
  Measured in mg/(kg*min)
AUCGIR,150-168h,SS - Area under the glucose infusion rate-time curve at steady state | From 150 to 168 hours after trial product administration (day 57)
  Measured in mg/kg
GIRmax,150-168h,SS - Maximum observed glucose infusion rate at steady state | From 150 to 168 hours after trial product administration (day 57)
  Measured in mg/(kg*min)
AUCGIR,0-24h,SS - Area under the glucose infusion rate-time curve at steady state | From 0 to 24 hours after trial product administration (day 14)
  Measured in mg/kg
GIRmax,0-24h,SS - Maximum observed glucose infusion rate at steady state | From 0 to 24 hours after trial product administration (day 14)
  Measured in mg/(kg*min)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Fukuoka, Japan

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com